CLINICAL TRIAL: NCT06324877
Title: Single Arm Open-label Clinical Trial in Ataxia-telangiectasia to Test the Effects of Nicotinamide Riboside on Ataxia Scales, Immune Function, and Neurofilament Light Chain.
Brief Title: Ataxia-telangiectasia: Treating Mitochondrial Dysfunction With Nicotinamide Riboside
Acronym: ATNAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HREC/24/QCHQ/106030
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-02

CONDITIONS: Ataxia Telangiectasia
Keywords: Dyskinesias; Neurologic Manifestations; Nervous System Diseases; Cerebellar Diseases; Brain Diseases; Central Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases; Spinocerebellar Ataxias; Neurocutaneous Syndromes; Genetic Diseases, Inborn; Primary Immunodeficiency Diseases; DNA Repair-Deficiency Disorders; Metabolic Diseases; Immunologic Deficiency Syndromes; Immune System Diseases; Ataxia; Cerebellar Ataxia; Ataxia Telangiectasia; Telangiectasis
MeSH Terms: conditions — Ataxia Telangiectasia; Dyskinesias; Neurologic Manifestations; Nervous System Diseases; Cerebellar Diseases; Brain Diseases; Central Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases; Spinocerebellar Ataxias; Neurocutaneous Syndromes; Genetic Diseases, Inborn; Primary Immunodeficiency Diseases; DNA Repair-Deficiency Disorders; Metabolic Diseases; Immunologic Deficiency Syndromes; Immune System Diseases; Ataxia; Cerebellar Ataxia; Telangiectasis | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: 1. Primary objective: Single arm open-label clinical trial in ataxia-telangiectasia to test the effects of nicotinamide riboside on ataxia scales, immune function, and neurofilament light chain.
  2. Secondary objectives:
     * Determine to what extent the beneficial effects ongoing of NR on NFl translate to clinical efficacy in patients with A-T.
     * Type 1 Interferon (INFs) epigenetic signature specifically the cGAS-STING pathway.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (full group) (Other): Single arm, open-label. Dose will be via oral capsule supplementation Nicotinamide Riboside at 25mg/kg/day divided into 3 doses (max 300mgs 3 times per day). Dosing will occur via 3 equal doses 3 times a day for 12 months.
  Interventions: Drug: Nicotinamide riboside

INTERVENTIONS:
Drug: Nicotinamide riboside — Oral capsule Nicotinamide Riboside 25mg/kg/day divided into 3 equal doses

SUMMARY:
Study design: Single arm open-label clinical trial in ataxia-telangiectasia to test the effects of nicotinamide riboside on ataxia scales, immune function, and neurofilament light chain. Study population: 6-10 patients with Ataxia-Telangiectasia. Dose: Nicotinamide riboside 25 mg/kg/day in 3 equal divided doses.

Primary endpoint: Scales for assessment and rating of ataxia (SARA), and International Cooperative Ataxia Rating Scale (ICARS). Improvement of at least ½ standard deviation in key clinical scales which includes either; a) significant improvement in total combined scores from the SARA and ICARS scales, and /or b) significant improvements any aspects of the SARA and ICARS scales individually, especially pertaining to; Postural and gait improvements, Improved syllable speed and articulation, Improved fine motor skills.

Secondary endpoints: Serum analysis of neurofilament light chain (Nfl), Type 1 Interferon (INFs) epigenetic signature

DETAILED DESCRIPTION:
Ataxia Telangiectasia (A-T) is a rare, genetic, progressive, life-limiting, neuro-degenerative condition affecting a variety of body systems resulting in ataxia, immune deficiency, respiratory complications and a predisposition to cancer. Currently there is no cure for A-T.

Over the years, a number of small clinical trials using steroids, antioxidants and anti-inflammatory agents have had little success. The disease natural history is relentless leading to early death. A-T generates a significant disease burden for the individuals, their extended families and on health care resources. With palliative care being the only current option for families, a treatment trial for A-T meets an unmet need. Our group previously demonstrated compelling evidence of reversible mitochondrial dysfunction and preventable cell death in A-T patient cells and the beneficial effects of heptanoate (C7), the primary metabolite of triheptanoin. C7 corrects a defect in endoplasmic reticulum (ER)-mitochondrial signalling in A-T cells and has great potential for application in treating patients. C7 has been utilised with efficacy and safety over the last 15 years for inborn errors of metabolism (IEM) such as long chain fatty acid defects (LC-FAOD).

A-T is due to a genetic defect that results in a defective serine/threonine protein kinase, known as ATM. Normally, ATM, plays a central role in protecting the genome against damage. It is increasingly evident that ATM protects cells against oxidative stress. This protein is also present outside the nucleus, where it is activated by oxidative stress through a separate mechanism from DNA damage, providing an explanation why anti-oxidants have a protective role in A-T cells in culture and in animal models. From these and other studies, it is evident that mitochondrial abnormalities characterise ATM and it has been suggested that A-T should be considered, at least in part, as a mitochondrial disease.

We have added substance to that claim by showing that ATM-deficient (B3) cells are exquisitely sensitive to inhibition of glycolysis by glucose deprivation, compared to controls (HBEC). We have also shown this increased sensitivity to nutrient deprivation for primary epithelial cells from patients and in immortalised patient cells. We demonstrated that this was caused by defective assembly of the VDAC1-GRP75-IP3R1 calcium channel and less ER-mitochondria contact points as determined by transmission electron microscopy. This in turn resulted in reduced calcium release from the ER and less transfer to mitochondria providing further evidence for mitochondrial dysfunction in A-T cells. We have recently completed a Phase 2A/B clinical trial exploring the efficacy and tolerability of C7 in AT patients (https://classic.clinicaltrials.gov/NCT04513002).

Nicotinamide adenine dinucleotide (NAD+) is an essential cofactor for many cellular enzymes, including those involved in mitochondrial biogenesis and maintenance. Nicotinamide adenine dinucleotide exists in two forms, including an oxidized (NAD+) and a reduced (NADH) form, and plays a key role in intermediary metabolism, as obligatory partner in numerous oxidation/reduction reactions. The cellular pool of NAD+ and NADH is tightly regulated through a careful balance between its biosynthesis and its breakdown by NAD+-consuming enzymes. NAD+ deficiency plays a role in disease mechanisms underlying DNA repair disorders. Mitochondrial damage and NAD+ depletion are key features in ataxia telangiectasia.

ATM-deficient mice have neuronal NAD+ deficiency, in particular in the cerebellum.

Fang et al. have demonstrated that mitochondrial dysfunction in ATM deficiency is linked to NAD+/SIRT1 inhibition. NAD+ replenishment significantly extends lifespan and improves health span in both ATM worms and mice through mitophagy and DNA repair. Treatments that replenish intracellular NAD+ reduce the severity of A-T neuropathology, normalize neuromuscular function, delay memory loss, and extend lifespan in both animal models. Mechanistically, treatments that increase intracellular NAD+ also stimulate neuronal DNA repair and improve mitochondrial quality via mitophagy.

Immune deficiency is common in AT, with most patients have humoral and cellular immune defects comprising immunoglobulin-A deficiency, immunoglobulin-G2 and immunoglobulin-G deficiency, and lymphopenia with low numbers of total and naive CD4 T cells. About 10% of patients with classic ataxia-telangiectasia present with hypogammaglobulinaemia with normal or raised immunoglobulin-M levels and follow a severe disease course. Recognition of foreign or misplaced nucleic acids is one of the principal modes by which the immune system detects pathogenic entities. When cytosolic DNA is sensed, a signal is relayed via the cGAS-STING pathway.

ATM deficient cells display elevated levels of INF- induced proteins, a feature also reported in sera of A-T patients. A double knockout of ATM and STING genes in mice attenuated autoinflammatory phenotypes, which was further decreased when the cGAS gene is also deleted in these mice. Inhibition of the cGAS-STING pathway ameliorates the premature senescence phenotype in AT brain organoids. Similar inflammatory manifestations are seen in patients with STING-associated vasculopathy in infancy which is an autosomal dominant type 1 interferonopathy.

Two groups have explored Nicotinamide Riboside (NR) supplementation in small groups of A-T patients via single arm, open label access, proof-of-concept clinical trials. Both have demonstrated improvements in validated ataxia scales. Improvements in immunoglobulin-G (IgG) levels were observed, no alterations were noted in NFlc. Improvements were lost in the wash out period. NR was well tolerated with no reported adverse events.

This is a single arm open-label clinical trial in ataxia-telangiectasia to test the effects of nicotinamide riboside on ataxia scales, immune function, and neurofilament light chain.

Dose will be via oral capsule supplementation at 25mg/kg/day divided into 3 doses (max 300mgs 3 times per day). Dosing will occur via 3 equal doses 3 times a day.

Primary efficacy endpoint: Improvement of at least ½ standard deviation in key clinical scales which includes either; a) significant improvement in total combined scores from the SARA and ICARS scales, and /or b) significant improvements any aspects of the SARA and ICARS scales individually, especially pertaining to; Postural and gait improvements, Improved syllable speed and articulation, Improved fine motor skills.

Secondary endpoints include: Serum analysis of neurofilament light chain (Nfl). Type 1 Interferon (INFs) epigenetic signature specifically the cGAS-STING pathway.

Safety endpoints: Treatment-related adverse events, Routine haematology and biochemical analyses, Paediatric Epilepsy Side Effects Questionnaire (PESQ), Regular clinical assessments.

ELIGIBILITY:
Inclusion Criteria:

Participants who meet all of the following criteria are eligible for enrolment:

* Patients of either sex, of any age, with a confirmed diagnosis of A-T,
* Patients who are able to undertake the study procedures,
* Families who are able to comply with the protocol for its duration and who provide informed patient assent and consent signed and dated by parent/legal guardian or adult participant according to local regulations.

Exclusion Criteria:

Participants who meet any of these criteria are not eligible for enrolment:

* Patients whose parents/legal guardians are not able to provide consent
* Patients who have been in another randomised clinical intervention trial where the use of investigational medicinal product within 3 months or 5 half-lives, whichever is longer, before study enrolment
* Taking off label mediations or nutritional supplements that the PI consider would impact participant's safe participation.
* Patients who are pregnant and/or lactating, planning a pregnancy during the study. Contraception must be used for sexually active male and female participants
* Liver enzymes (alanine aminotransferase [ALT]/aspartate aminotransferase [AST]) or total bilirubin > 2 x the upper limit of normal at the time of screening.
* Renal insufficiency as defined by estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2 at the screening visit.
* Any comorbid medical condition that in the assessment of the PI that would impact participant's safe participation (e.g. active cancer requiring treatment)
* Evidence of dysphagia that places subject at risk of aspiration if orally fed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Scales for assessment and rating of ataxia | 4 monthly assessment over 12 months
  Scales for assessment and rating of ataxia is a validated cerebellar ataxia tool, measuring gait (scale 0-8), stance (scale 0-6), sitting (scale 0-4), speech (scale 0-6), finger-chase test scale 0-4), finger nose-test (scale 0-4), fast alternating movements (scale 0-4) and heel-shin test (scale 0-4). 0 indicates normal function, escalating numbers in the scale domains indicate increased difficultly with the measured tasks.
International Cooperative Ataxia Rating Scale | 4 monthly assessment over 12 months
  International Cooperative Ataxia Rating Scale is a scale recorded out of 100 with 19 items and 4 sub-scales and has been used in A-T. 0 indicates normal function, escalating numbers in the scale domains indicate increased difficulty with the measured tasks.

SECONDARY OUTCOMES:
Serum analysis of neurofilament light chain | 12 months
  Neurofilament light chain (Nfl) will be quantified using the single-molecule (Simoa) array method and the Simoa NF-light assay (Quanterix, MA, US) on an HD-1platform (GBIO). Levels of neurofilament light chain will be correlated with clinical endpoints.
Type 1 Interferon epigenetic signature | 12 months
  An IFN signature will be investigated by measuring six IFN-stimulated genes (ISGs) by quantitative PCR (QPCR).

OTHER OUTCOMES:
Quality of Life Measures | 4 monthly assessment over 12 months
  Paediatric Side Effect Questionnaire is a 19-item measure consisting of five sub-scales: cognitive (six items), motor (four items), behavioural (three items), general neurological (four items), and weight (two items) side effects. The investigators will add five items for gastrointestinal side effects to the questionnaire, including gastrointestinal pain, acid reflux, vomiting, diarrhoea, and constipation. The scale will be recorded from 0 to 96. 0 indicates normal function, escalating numbers in the scale domains indicate increased difficultly with the measured task.

CONTACTS AND LOCATIONS:
Overall Officials: David Coman, MBBS FRACP, Principal Investigator — Queensland Children's Hospital
Locations (1):
- Queensland Children's Hospital, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Veenhuis SJG, van Os NJH, Janssen AJWM, van Gerven MHJC, Coene KLM, Engelke UFH, Wevers RA, Tinnevelt GH, Ter Heine R, van de Warrenburg BPC, Weemaes CMR, Roeleveld N, Willemsen MAAP. Nicotinamide Riboside Improves Ataxia Scores and Immunoglobulin Levels in Ataxia Telangiectasia. Mov Disord. 2021 Dec;36(12):2951-2957. doi: 10.1002/mds.28788. Epub 2021 Sep 13. PMID 34515380
- [Background] Fang EF, Kassahun H, Croteau DL, Scheibye-Knudsen M, Marosi K, Lu H, Shamanna RA, Kalyanasundaram S, Bollineni RC, Wilson MA, Iser WB, Wollman BN, Morevati M, Li J, Kerr JS, Lu Q, Waltz TB, Tian J, Sinclair DA, Mattson MP, Nilsen H, Bohr VA. NAD+ Replenishment Improves Lifespan and Healthspan in Ataxia Telangiectasia Models via Mitophagy and DNA Repair. Cell Metab. 2016 Oct 11;24(4):566-581. doi: 10.1016/j.cmet.2016.09.004. PMID 27732836
- [Background] Zannolli R, Buoni S, Betti G, Salvucci S, Plebani A, Soresina A, Pietrogrande MC, Martino S, Leuzzi V, Finocchi A, Micheli R, Rossi LN, Brusco A, Misiani F, Fois A, Hayek J, Kelly C, Chessa L. A randomized trial of oral betamethasone to reduce ataxia symptoms in ataxia telangiectasia. Mov Disord. 2012 Sep 1;27(10):1312-6. doi: 10.1002/mds.25126. Epub 2012 Aug 23. PMID 22927201
- [Background] Woelke S, Pommerening H, Kieslich M, Schubert R, Zielen S. Growth hormone treatment in patients with ataxia telangiectasia. Growth Factors. 2017 Jun;35(2-3):125-130. doi: 10.1080/08977194.2017.1367681. PMID 28948852
- [Background] Chessa L, Leuzzi V, Plebani A, Soresina A, Micheli R, D'Agnano D, Venturi T, Molinaro A, Fazzi E, Marini M, Ferremi Leali P, Quinti I, Cavaliere FM, Girelli G, Pietrogrande MC, Finocchi A, Tabolli S, Abeni D, Magnani M. Intra-erythrocyte infusion of dexamethasone reduces neurological symptoms in ataxia teleangiectasia patients: results of a phase 2 trial. Orphanet J Rare Dis. 2014 Jan 9;9:5. doi: 10.1186/1750-1172-9-5. PMID 24405665
- [Background] Nissenkorn A, Borgohain R, Micheli R, Leuzzi V, Hegde AU, Mridula KR, Molinaro A, D'Agnano D, Yareeda S, Ben-Zeev B. Development of global rating instruments for pediatric patients with ataxia telangiectasia. Eur J Paediatr Neurol. 2016 Jan;20(1):140-6. doi: 10.1016/j.ejpn.2015.09.002. Epub 2015 Sep 25. PMID 26493850
- [Background] Airhart SE, Shireman LM, Risler LJ, Anderson GD, Nagana Gowda GA, Raftery D, Tian R, Shen DD, O'Brien KD. An open-label, non-randomized study of the pharmacokinetics of the nutritional supplement nicotinamide riboside (NR) and its effects on blood NAD+ levels in healthy volunteers. PLoS One. 2017 Dec 6;12(12):e0186459. doi: 10.1371/journal.pone.0186459. eCollection 2017. PMID 29211728
- [Background] Chen P, Peng C, Luff J, Spring K, Watters D, Bottle S, Furuya S, Lavin MF. Oxidative stress is responsible for deficient survival and dendritogenesis in purkinje neurons from ataxia-telangiectasia mutated mutant mice. J Neurosci. 2003 Dec 10;23(36):11453-60. doi: 10.1523/JNEUROSCI.23-36-11453.2003. PMID 14673010
- [Background] Paap BK, Roeske S, Durr A, Schols L, Ashizawa T, Boesch S, Bunn LM, Delatycki MB, Giunti P, Lehericy S, Mariotti C, Melegh J, Pandolfo M, Tallaksen CME, Timmann D, Tsuji S, Schulz JB, van de Warrenburg BP, Klockgether T. Standardized Assessment of Hereditary Ataxia Patients in Clinical Studies. Mov Disord Clin Pract. 2016 Feb 11;3(3):230-240. doi: 10.1002/mdc3.12315. eCollection 2016 May-Jun. PMID 30363623
- [Background] Gueven N, Luff J, Peng C, Hosokawa K, Bottle SE, Lavin MF. Dramatic extension of tumor latency and correction of neurobehavioral phenotype in Atm-mutant mice with a nitroxide antioxidant. Free Radic Biol Med. 2006 Sep 15;41(6):992-1000. doi: 10.1016/j.freeradbiomed.2006.06.018. Epub 2006 Jul 4. PMID 16934683
- [Background] Guo Z, Kozlov S, Lavin MF, Person MD, Paull TT. ATM activation by oxidative stress. Science. 2010 Oct 22;330(6003):517-21. doi: 10.1126/science.1192912. PMID 20966255
- [Background] Valentin-Vega YA, Maclean KH, Tait-Mulder J, Milasta S, Steeves M, Dorsey FC, Cleveland JL, Green DR, Kastan MB. Mitochondrial dysfunction in ataxia-telangiectasia. Blood. 2012 Feb 9;119(6):1490-500. doi: 10.1182/blood-2011-08-373639. Epub 2011 Dec 5. PMID 22144182
- [Background] Yeo AJ, Chong KL, Gatei M, Zou D, Stewart R, Withey S, Wolvetang E, Parton RG, Brown AD, Kastan MB, Coman D, Lavin MF. Impaired endoplasmic reticulum-mitochondrial signaling in ataxia-telangiectasia. iScience. 2020 Dec 23;24(1):101972. doi: 10.1016/j.isci.2020.101972. eCollection 2021 Jan 22. PMID 33437944
- [Background] Lautrup S, Sinclair DA, Mattson MP, Fang EF. NAD+ in Brain Aging and Neurodegenerative Disorders. Cell Metab. 2019 Oct 1;30(4):630-655. doi: 10.1016/j.cmet.2019.09.001. PMID 31577933
- [Background] Zapata-Perez R, Wanders RJA, van Karnebeek CDM, Houtkooper RH. NAD+ homeostasis in human health and disease. EMBO Mol Med. 2021 Jul 7;13(7):e13943. doi: 10.15252/emmm.202113943. Epub 2021 May 27. PMID 34041853
- [Background] Subramanian GN, Yeo AJ, Gatei MH, Coman DJ, Lavin MF. Metabolic Stress and Mitochondrial Dysfunction in Ataxia-Telangiectasia. Antioxidants (Basel). 2022 Mar 28;11(4):653. doi: 10.3390/antiox11040653. PMID 35453338
- [Background] Stern N, Hochman A, Zemach N, Weizman N, Hammel I, Shiloh Y, Rotman G, Barzilai A. Accumulation of DNA damage and reduced levels of nicotine adenine dinucleotide in the brains of Atm-deficient mice. J Biol Chem. 2002 Jan 4;277(1):602-8. doi: 10.1074/jbc.M106798200. Epub 2001 Oct 25. PMID 11679583
- [Background] Yang B, Dan X, Hou Y, Lee JH, Wechter N, Krishnamurthy S, Kimura R, Babbar M, Demarest T, McDevitt R, Zhang S, Zhang Y, Mattson MP, Croteau DL, Bohr VA. NAD+ supplementation prevents STING-induced senescence in ataxia telangiectasia by improving mitophagy. Aging Cell. 2021 Apr;20(4):e13329. doi: 10.1111/acel.13329. Epub 2021 Mar 18. PMID 33734555
- [Background] Aguado J, Chaggar HK, Gomez-Inclan C, Shaker MR, Leeson HC, Mackay-Sim A, Wolvetang EJ. Inhibition of the cGAS-STING pathway ameliorates the premature senescence hallmarks of Ataxia-Telangiectasia brain organoids. Aging Cell. 2021 Sep;20(9):e13468. doi: 10.1111/acel.13468. Epub 2021 Aug 30. PMID 34459078
- [Background] Presterud R, Deng WH, Wennerstrom AB, Burgers T, Gajera B, Mattsson K, Solberg A, Fang EF, Nieminen AI, Stray-Pedersen A, Nilsen H. Long-Term Nicotinamide Riboside Use Improves Coordination and Eye Movements in Ataxia Telangiectasia. Mov Disord. 2024 Feb;39(2):360-369. doi: 10.1002/mds.29645. Epub 2023 Oct 29. PMID 37899683
- [Background] van Os NJH, Jansen AFM, van Deuren M, Haraldsson A, van Driel NTM, Etzioni A, van der Flier M, Haaxma CA, Morio T, Rawat A, Schoenaker MHD, Soresina A, Taylor AMR, van de Warrenburg BPC, Weemaes CMR, Roeleveld N, Willemsen MAAP. Ataxia-telangiectasia: Immunodeficiency and survival. Clin Immunol. 2017 May;178:45-55. doi: 10.1016/j.clim.2017.01.009. Epub 2017 Jan 24. PMID 28126470
- [Background] Kim J, Gupta R, Blanco LP, Yang S, Shteinfer-Kuzmine A, Wang K, Zhu J, Yoon HE, Wang X, Kerkhofs M, Kang H, Brown AL, Park SJ, Xu X, Zandee van Rilland E, Kim MK, Cohen JI, Kaplan MJ, Shoshan-Barmatz V, Chung JH. VDAC oligomers form mitochondrial pores to release mtDNA fragments and promote lupus-like disease. Science. 2019 Dec 20;366(6472):1531-1536. doi: 10.1126/science.aav4011. Epub 2019 Dec 19. PMID 31857488
- [Background] Gul E, Sayar EH, Gungor B, Eroglu FK, Surucu N, Keles S, Guner SN, Findik S, Alpdundar E, Ayanoglu IC, Kayaoglu B, Geckin BN, Sanli HA, Kahraman T, Yakicier C, Muftuoglu M, Oguz B, Cagdas Ayvaz DN, Gursel I, Ozen S, Reisli I, Gursel M. Type I IFN-related NETosis in ataxia telangiectasia and Artemis deficiency. J Allergy Clin Immunol. 2018 Jul;142(1):246-257. doi: 10.1016/j.jaci.2017.10.030. Epub 2017 Nov 16. PMID 29155101
- [Background] Siddoo-Atwal C, Haas AL, Rosin MP. Elevation of interferon beta-inducible proteins in ataxia telangiectasia cells. Cancer Res. 1996 Feb 1;56(3):443-7. PMID 8564949
- [Background] Hartlova A, Erttmann SF, Raffi FA, Schmalz AM, Resch U, Anugula S, Lienenklaus S, Nilsson LM, Kroger A, Nilsson JA, Ek T, Weiss S, Gekara NO. DNA damage primes the type I interferon system via the cytosolic DNA sensor STING to promote anti-microbial innate immunity. Immunity. 2015 Feb 17;42(2):332-343. doi: 10.1016/j.immuni.2015.01.012. PMID 25692705
- [Background] Song X, Ma F, Herrup K. Accumulation of Cytoplasmic DNA Due to ATM Deficiency Activates the Microglial Viral Response System with Neurotoxic Consequences. J Neurosci. 2019 Aug 7;39(32):6378-6394. doi: 10.1523/JNEUROSCI.0774-19.2019. Epub 2019 Jun 12. PMID 31189575
- [Background] Paul BD, Snyder SH, Bohr VA. Signaling by cGAS-STING in Neurodegeneration, Neuroinflammation, and Aging. Trends Neurosci. 2021 Feb;44(2):83-96. doi: 10.1016/j.tins.2020.10.008. Epub 2020 Nov 10. PMID 33187730